CLINICAL TRIAL: NCT07258251
Title: Strengthening Hepatitis B Screening, Linkage to Care and Long-Term Monitoring in Phichit Province, Thailand: A Birth Bohort Approach
Acronym: HBV-PHICHIT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Task Force for Global Health (Other)
Collaborators: Phichit Provincial Public Health Office, Ministry of Public Health, Thailand (Host institution) (Unknown); Division of Gastroenterology, Department of Medicine Siriraj Hospital, Mahidol University (Unknown); Ministry of Health, Thailand (Other Government); Phichit Provincial Hospital (Unknown); Liver Foundation Thailand (Unknown); Thai Association for the Study of the Liver (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC102_68BT-MED35_COR-HEPB
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Hepatitis B; Hepatitis B Virus Infection
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implementation Cohort (Experimental): Implementation Cohort (Single Arm)
  Interventions:
  1. Drug: Tenofovir Alafenamide (TAF) HBsAg-positive individuals meeting WHO 2024 treatment eligibility criteria will receive daily oral TAF. Tenofovir disoproxil fumarate (TDF) may be used if TAF is unavailable.
  2. Behavioral: Community-Based Support Interventions to improve linkage to care, retention, and treatment adherence4646. This includes telephone calls, home visits by community health volunteers, and phone/SMS reminders for appointments.
  3. Diagnostic Test: Simplified WHO 2024 Criteria HBsAg-positive individuals will be evaluated for treatment eligibility using simplified 2024 WHO guidelines, including APRI score, as an alternative to HBV DNA testing.
  Interventions: Drug: Tenofovir Alafenamide (TAF); Behavioral: Community-Based Support; Diagnostic Test: Simplified WHO 2024 Criteria

INTERVENTIONS:
Drug: Tenofovir Alafenamide (TAF) — HBsAg-positive individuals meeting WHO 2024 treatment eligibility criteria will receive daily oral TAF. Tenofovir disoproxil fumarate (TDF) may be used if TAF is unavailable.
Behavioral: Community-Based Support — Interventions to improve linkage to care, retention, and treatment adherence. This includes telephone calls, home visits by community health volunteers, and phone/SMS reminders for appointments.
Diagnostic Test: Simplified WHO 2024 Criteria — HBsAg-positive individuals will be evaluated for treatment eligibility using simplified 2024 WHO guidelines, including APRI score, as an alternative to HBV DNA testing.

SUMMARY:
This study in Phichit province, Thailand, aims to find and support adults born before 1992 who are at high risk for hepatitis B infection. Many people in this group were born before the universal hepatitis B vaccine was available and may not know they are infected. The study will invite nearly 240,000 eligible adults for free hepatitis B screening. Those who test positive will be linked to care at one of 12 district hospitals. Doctors will use simplified 2024 World Health Organization (WHO) guidelines to decide who needs treatment. Eligible individuals will receive a safe, effective daily medicine (tenofovir alafenamide). The study will use community health volunteers and phone reminders to help patients stay in care and take their medication regularly. Over three years, the study will track improvements in liver health and virus levels, aiming to prevent liver cirrhosis and cancer.

DETAILED DESCRIPTION:
Chronic hepatitis B virus (HBV) infection is a significant cause of liver cirrhosis and hepatocellular carcinoma (HCC) in Thailand. While Thailand's universal infant vaccination program, implemented in 1992, has been successful, adults born before this date remain a high-risk population with an estimated 2-3 million chronic infections.

Despite free access to HBsAg screening and treatment (including TAF/TDF), barriers such as the lack of reimbursement for HBV DNA testing and poor linkage to care have hampered progress toward WHO 2030 elimination targets.

This study is a pragmatic implementation research project designed to scale up HBsAg screening, linkage to care, and long-term monitoring in Phichit Province. It targets the birth cohort of adults born before 1992 (approx. 238,786 people).

The study will develop and evaluate tools to identify unscreened individuals, improve linkage to dedicated viral hepatitis clinics, and support long-term adherence. A key component is the implementation of simplified WHO 2024 treatment criteria, which utilize non-invasive markers like the APRI score as an alternative to HBV DNA testing to determine treatment eligibility.

ELIGIBILITY:
Inclusion Criteria:

* Adults born before January 1, 1992
* Residing in Phichit Province
* Individuals who test positive for HBsAg will be invited to participate in the follow-up cohort
* HBsAg positive patients who are already under care will also be invited to participate

Exclusion Criteria:

* Subjects who withdraw consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
HBsAg Screening Uptake | 36 months
  Percentage of the target population (adults born before Jan
  1, 1992, in Phichit province) who are successfully screened for HBsAg. (Target: 90%)
Linkage to Care | 36 months
  Percentage of individuals who test positive for HBsAg and are successfully linked to care for clinical assessment and treatment evaluation.
Treatment Initiation | 36 months
  Percentage of HBsAg-positive individuals identified as eligible for treatment (per WHO 2024 guidelines) who successfully initiate antiviral therapy

SECONDARY OUTCOMES:
Treatment Eligibility (Simplified Criteria) | 36 months
  Proportion of HBsAg-positive individuals eligible for treatment based on simplified WHO 2024 criteria without HBV DNA results (e.g., using APRI score)
Treatment Adherence | 12 Months and 24 Months
  Proportion of patients on treatment with good compliance, defined as taking & 80% of prescribed medication, measured by pill count and the 8-item Morisky Medication Adherence Scale (MMAS-8)
Retention in Care | 12 Months, 24 Months, and 36 Months
  Proportion of all HBsAg-positive individuals (treated and untreated) who maintain scheduled 6-monthly follow-up appointments.
Effectiveness of Community-Based Support | 36 Months
  Assessed by measuring the impact of iinterventions (e.g., health volunteers, phone reminders) on linkage and retention rates
Virologic Response | Baseline, 12 Months, 24 Months, 36 Months
  Change in HBV DNA viral load from baseline among treated patients
Biochemical Response | Baseline and every 6 months for 36 months
  Proportion of treated patients achieving ALT normalization
Fibrosis/Inflammation Response | Baseline and every 6 months for 36 months
  Change in APRI score from baseline among treated patients
HBsAg Serometrics | Baseline, 12 Months, 24 Months, 36 Months
  Change in quantitative HBsAg (qHBsAg) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Professor Tawasek Tawandee, Principal Investigator — Mahidol University
Locations (1):
- Phichit Provincial Hospital, Phichit / 12 District Hospitals in Phichit Province, Phichit, Changwat Phichit, Thailand